CLINICAL TRIAL: NCT04901845
Title: VEIN Health Chronic Venous Disease at Primary and Specialized Healthcare Level -Update on Prevalence and Characteristics
Brief Title: VEIN Health - CVD Prevalence and Characteristics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bokhua Memorial Cardiovascular Center (Other)
Collaborators: Chapidze Emergency Cardiology Center (Unknown)
Responsible Party: Principal Investigator, Mamuka Bokuchava, TSSU Professor; Deputy Director of Bokhua Memorial Cardiovascular Center, Bokhua Memorial Cardiovascular Center
Other Study IDs: IC4-05682-009-GEO
Record Dates: First submitted 2021-05-05; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Chronic Venous Disease
Keywords: Chronic Venous Disease; Prevalence; Characteristics; Management tactics evaluation; Risk-factors; Distribution of CEAP stages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients applying to Primary Healthcare Consultation: Consequent patients applying to the Primary healthcare to consult for any reason during 2 week period
  Interventions: Other: No intervention provided
- Patients applying to Specialized Healthcare Consultation: Consequent patients applying to the Specialized healthcare to consult for any reason during 2 week period
  Interventions: Other: No intervention provided

INTERVENTIONS:
Other: No intervention provided — Study is provided in the usual daily practice of the physicians without interventions made in their practice

SUMMARY:
Epidemiology Study to learn prevalence and characteristics of CVD at Primary and Specialized healthcare level

DETAILED DESCRIPTION:
Cross sectional study that will evaluate prevalence, characteristics, diagnostic and treatment status of the patients with Chronic Venous Disease at primary or specialized healthcare level during 2 week period. No interventions are made. Information on patient demographic, physical, clinical parameters, medical history data and procedures performed during visit in routine daily practice of physicians is registered and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Patient consented to participate

Exclusion Criteria:

* Patient applying due to emergency situation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients applying to consultation due to any reason
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Prevalence of CVD | 2 weeks
  Percent of CVD symptomatic patients among patients applying to consultation for any reason
Distribution of CEAP stages | 2 weeks
  Percent of CVD patients with various CEAP stages
Prevalence of risk-factors associated with CVD | 2 weeks
  Frequency of risk-factors associated with CVD
Management tactics | 2 weeks
  Tactics chosen by physicians to manage CVD

CONTACTS AND LOCATIONS:
Overall Officials: Nugzar Pargalava, MD, PhD, Study Director — Bokhua Memorial Cardiovascular Center; Zaza Lazarahvili, MD, PhD, Study Director — Chapidze Emergency Cardiology Center; Mamuka Bokuchava, MD, PhD, Study Director — Bokhua Memorial Cardiovascular Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shabani Varaki E, Gargiulo GD, Penkala S, Breen PP. Peripheral vascular disease assessment in the lower limb: a review of current and emerging non-invasive diagnostic methods. Biomed Eng Online. 2018 May 11;17(1):61. doi: 10.1186/s12938-018-0494-4. PMID 29751811
- [Background] Nicolaides A, Kakkos S, Baekgaard N, Comerota A, de Maeseneer M, Eklof B, Giannoukas AD, Lugli M, Maleti O, Myers K, Nelzen O, Partsch H, Perrin M. Management of chronic venous disorders of the lower limbs. Guidelines According to Scientific Evidence. Part I. Int Angiol. 2018 Jun;37(3):181-254. doi: 10.23736/S0392-9590.18.03999-8. No abstract available. PMID 29871479
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] Rabe E, Guex JJ, Puskas A, Scuderi A, Fernandez Quesada F; VCP Coordinators. Epidemiology of chronic venous disorders in geographically diverse populations: results from the Vein Consult Program. Int Angiol. 2012 Apr;31(2):105-15. PMID 22466974